CLINICAL TRIAL: NCT02826785
Title: Feasibility and Optimization of a Cognitive Intervention for Parkinson Disease
Acronym: FOCI-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Erin Foster, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201403072
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive strategy training (Experimental): The cognitive strategy training intervention consists of 6 weekly ~1 hour sessions. It is delivered in an individual, face-to-face format in the client's home. It is a behavioral intervention that teaches people metacognitive, problem-solving and other compensatory strategies to address self-identified cognitive performance problems, and it uses practice and homework to promote strategy learning, retention and transfer.
  Interventions: Behavioral: Cognitive strategy training

INTERVENTIONS:
Behavioral: Cognitive strategy training — The intervention teaches strategies in a way that promotes generalization and enhances daily function . It includes four core elements known to enhance learning transfer: (1) self-generation of broadly applicable strategies, (2) practice across multiple contexts and activities, (3) emphasis on metacognition, and (4) use of meaningful everyday activities.

SUMMARY:
This study investigates the feasibility of a cognitive strategy training intervention for people with Parkinson disease (PD). We plan to recruit 8 non-demented PD participants to complete 6 weekly treatment sessions and Pre- and Post-testing (8 sessions total, entire study duration per participant = 8 weeks). We will measure participant responsiveness and the overall efficiency of the intervention process.

DETAILED DESCRIPTION:
Cognitive impairment is common in Parkinson disease (PD) and is a significant source of disability and reduced quality of life. Existing rehabilitative interventions, which focus on cognitive process training, have not been successful in mitigating its negative functional consequences. We have developed a client-centered cognitive strategy training intervention to enable people with PD to work around their cognitive deficits and maintain their functional performance. This study is an exploratory case series to assess aspects of its feasibility. Specifically, we will assess participant responsiveness to the intervention (acceptance, engagement, adherence), and we will track logistical information (e.g., scheduling). We will also administer an exploratory outcome measure of treatment effect to gain preliminary evidence on the effect of the intervention on self-identified cognitive performance problems. This information will guide modifications and enhancements in preparation for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over age 50 who meet criteria for idiopathic typical PD, are Hoehn & Yahr stage I-III (mild to moderate disease; Hoehn & Yahr, 1967) and are treated with levodopa/carbidopa. For this early phase of development we will limit enrollment to people who can identify at least one daily cognitive performance problem and are willing to learn strategies to address it.

Exclusion Criteria:

* Possible dementia, medication change over the study period, other neurological disorders, brain surgery (e.g., STN DBS), history of psychotic disorder or significant current psychiatric disorder (i.e., moderate to severe anxiety, apathy or depression), or any condition that would interfere with participation (e.g., non-English speaking). Participants taking benzos will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erin R Foster, PhD, Principal Investigator — Washington University School of Medicine